CLINICAL TRIAL: NCT07293702
Title: **Effect of Instrument-Assisted Soft Tissue Mobilization on Pain, Functionality, and Proprioception in Individuals With Subacromial Impingement Syndrome**
Brief Title: IASTM Effects on Pain, Functionality, and Proprioception in Subacromial Impingement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-6969
Record Dates: First submitted 2025-12-01; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Subacromial Impingement Syndrome; Massage; Instrument-Assisted Soft Tissue Mobilization; Soft Tissue Injuries
Keywords: Subakromial Impingement Syndrome; IASTM; Shoulder
MeSH Terms: conditions — Shoulder Impingement Syndrome; Soft Tissue Injuries

STUDY DESIGN:
Intervention Model Description: Participants in the first group underwent conventional physiotherapy interventions for 4 weeks, 3 days per week.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional exercise group (Active Comparator): Conventional exercises will be applied.
  Interventions: Other: Conventional exercise group
- IASTM group (Experimental): In addition to the conventional exercises, Instrument-Assisted Soft Tissue Mobilization (IASTM) will be applied.
  Interventions: Other: Conventional exercise group; Other: IASTM group

INTERVENTIONS:
Other: Conventional exercise group — All participants will receive a standardized electrotherapy program in a clinical setting, consisting of TENS (100 Hz, 30 minutes), ultrasound (1.5 W/cm², 8 minutes), and a 15-minute cold-pack application, delivered three times per week for four weeks. In addition to electrotherapy, participants in the conventional exercise group will perform a physiotherapist-guided exercise program aimed at improving shoulder flexion, abduction, internal and external rotation through stretching and range-of-motion exercises. The program will include Codman exercises, wand exercises, finger-ladder activities, and condition-appropriate strengthening exercises, progressed according to each participant's pain level and tolerance.
Other: IASTM group — Participants in the IASTM group will receive Instrument-Assisted Soft Tissue Mobilization in addition to the conventional treatment program, three days per week for four weeks, for a total of 12 sessions. The IASTM technique will be applied to the subscapularis, anterior deltoid, biceps brachii, upper trapezius, supraspinatus, infraspinatus, teres major, teres minor, and posterior deltoid muscles.
  For each muscle group, the treatment will be administered for 20 seconds in a parallel direction and 20 seconds in a perpendicular direction, using sweep and brush techniques at an angle of approximately 45 degrees.
  Arms: IASTM group

SUMMARY:
The aim of this study will be to investigate the effects of Instrument-Assisted Soft Tissue Mobilization (IASTM), applied in addition to a conventional exercise program, on pain, range of motion, proprioception, functionality, and quality of life in individuals with Subacromial Impingement Syndrome (SIS).

DETAILED DESCRIPTION:
The aim of this study will be to investigate the effects of Instrument-Assisted Soft Tissue Mobilization (IASTM), applied in addition to a conventional exercise program, on pain, range of motion, proprioception, functionality, and quality of life in individuals with Subacromial Impingement Syndrome (SIS).

A total of 38 participants will be included in the study and will be randomly assigned to either the Conventional Exercise Group or the IASTM Group. Both groups will receive treatment for 4 weeks, three sessions per week, for a total of 12 sessions.

Before the intervention, both groups will be assessed for pain (VAS), range of motion (goniometer), joint position sense (goniometer), functionality (Disabilities of the Arm, Shoulder and Hand - DASH), and quality of life (Rotator Cuff Quality of Life - RC-QoL).

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with SIS by MRI
* Men and women between 40 and 60 years of age
* Individuals with symptoms persisting for at least one month
* Individuals with a minimum of 60° of shoulder flexion and abduction range of motion

Exclusion Criteria:

* Individuals with a history of surgery on the affected arm
* Individuals with an open wound on the arm
* Individuals with an active infection
* Individuals with inflammatory joint disease
* Individuals with malignant or benign tumors were excluded from the study.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | From enrollment to the end of treatment at 4 weeks
  The Visual Analog Scale (VAS) is a tool used to measure pain intensity as a single-dimensional construct across different adult populations. It typically consists of a horizontal or vertical line measuring 10 cm in length. On this scale, a score of 0 indicates no pain, while a score of 10 represents the worst pain imaginable.
Range of motion | From enrollment to the end of treatment at 4 weeks
  Shoulder flexion, abduction, internal rotation, and external rotation range of motion will be assessed using a universal goniometer while the patient is positioned in supine and performs the movements actively.
The Disabilities of the Arm, Shoulder and Hand (DASH) | From enrollment to the end of treatment at 4 weeks
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire is a scale that evaluates functional status and capability following injuries or disorders affecting the upper extremity. The DASH consists of 30 items. These items assess difficulties encountered during specific tasks, as well as pain, numbness, stiffness, weakness, sleep problems, self-confidence, and participation in social activities. Scores range from 0 to 100, with higher scores indicating greater impairment in upper extremity function.

SECONDARY OUTCOMES:
Joint position sense | From enrollment to the end of treatment at 4 weeks
  To evaluate shoulder proprioception, joint position sense will be measured at 60° of shoulder flexion and 60° of shoulder abduction. During the assessment, participants will be positioned in standing and guided to the target angles by the physiotherapist using a goniometer. In each position, participants will be asked to maintain 60° of flexion or 60° of abduction for 10 seconds with their eyes open and to memorize the perceived position. They will then be instructed to reproduce the same movement with their eyes closed. The difference between the angle measured with eyes open and the angle reproduced with eyes closed will be recorded as the joint position sense error (error angle).
Rotator cuff quality of life Index | From enrollment to the end of treatment at 4 weeks
  Quality of life in individuals with shoulder pathology was evaluated using the Rotator Cuff Quality of Life (RC-QoL) questionnaire. The RC-QoL consists of 34 items and five subscales. Results are interpreted in a positive direction; as the RC-QoL score increases, the individual's shoulder-related quality of life is considered to have improved, and symptoms are regarded as reduced.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, PhD, Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No